CLINICAL TRIAL: NCT00369941
Title: A Multicenter, Double-Blind, Randomized, Active-Controlled Study to Evaluate the Safety and Antiretroviral Activity of MK-0518 Versus Efavirenz in Treatment Naive HIV-Infected Patients, Each in Combination With TRUVADA™
Brief Title: A Study to Evaluate the Safety and Antiretroviral Activity of MK-0518 Versus Efavirenz in Treatment Naive HIV-Infected Patients, Each in Combination With TRUVADA (0518-021 EXT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0518-021; MK-0518-021 (Other: Merck); 2006_519 (Other: Merck Registration ID)
Record Dates: First submitted 2006-08-29; First posted 2006-08-30 (Estimated); Results first posted 2010-05-11 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-0518 400 mg b.i.d. (Experimental): MK-0518 400 mg, which can be taken by mouth (PO) twice a day (b.i.d.) without regard to food, and placebo to efavirenz, which will be taken PO at bedtime (q.h.s.) on an empty stomach preferably at bedtime. All participants will take one tablet of TRUVADA® (200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate) with food, daily with the morning dose of MK-0518. Dosing interval adjustment of TRUVADA® is recommended in all participants with creatinine clearance 30-49 mL/min.
  Interventions: Drug: MK-0518; Drug: Comparator: Truvada; Drug: Comparator: Placebo to efavirenz
- Efavirenz 600 mg q.h.s. (Active Comparator): Efavirenz 600 mg, which will be taken by mouth (PO) at bedtime (q.h.s.) on an empty stomach preferably at bedtime, and placebo to MK-0518, which will be taken PO twice a day (b.i.d.) without regard to food. All participants will take one tablet of TRUVADA® with food, daily with the morning dose of placebo. Dosing interval adjustment of TRUVADA® is recommended in all participants with creatinine clearance 30-49 mL/min.
  Interventions: Drug: Comparator: efavirenz; Drug: Comparator: Truvada; Drug: Comparator: Placebo to MK-0518

INTERVENTIONS:
Drug: MK-0518 — 400 mg MK-0518 tablet taken by mouth (PO) twice a day (b.i.d.) for up to 240 weeks
  Other Names: raltegravir; Isentress®
  Arms: MK-0518 400 mg b.i.d.
Drug: Comparator: efavirenz — 600 mg efavirenz tablet taken by mouth (PO) every night (q.h.s.) for up to 240 weeks
  Other Names: Sustiva®
  Arms: Efavirenz 600 mg q.h.s.
Drug: Comparator: Truvada — One tablet Truvada once a day (q.d.) for up to 240 weeks (one tablet contains 200 mg emtricitabine and 300 mg tenofovir)
  Other Names: emtricitabine/tenofovir disoproxil fumarate
Drug: Comparator: Placebo to MK-0518 — Placebo to MK-0518 PO b.i.d., taken for up to 240 weeks
  Arms: Efavirenz 600 mg q.h.s.
Drug: Comparator: Placebo to efavirenz — Placebo to efavirenz PO every night (q.h.s.), taken for up to 240 weeks
  Arms: MK-0518 400 mg b.i.d.

SUMMARY:
This study will investigate the safety and efficacy of MK-0518 versus efavirenz, in combination with TRUVADA, as a therapy for Human Immunodeficiency Virus (HIV)-infected patients not previously treated.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a male or female at least 18 years of age
* Participant is HIV positive
* Participant is naïve to antiretroviral therapy (ART) and has not received any ART

Exclusion Criteria:

* Participant has received approved or experimental antiretroviral agents in the past
* Participant has been treated for a viral infection other than HIV such as hepatitis B virus infection with an agent that is active against HIV including but not limited to adefovir or lamivudine (= 7 days total)
* Participant has documented resistance to tenofovir, emtricitabine, and/or efavirenz
* Participant has used another experimental HIV-integrase inhibitor
* Participant has a current (active) diagnosis of acute hepatitis due to any cause
* Participants with chronic hepatitis including chronic hepatitis B and/or C may enter the study as long as they have stable liver function tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2006-08; Primary Completion 2009-05 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Lennox JL, DeJesus E, Lazzarin A, Pollard RB, Madruga JV, Berger DS, Zhao J, Xu X, Williams-Diaz A, Rodgers AJ, Barnard RJ, Miller MD, DiNubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK investigators. Safety and efficacy of raltegravir-based versus efavirenz-based combination therapy in treatment-naive patients with HIV-1 infection: a multicentre, double-blind randomised controlled trial. Lancet. 2009 Sep 5;374(9692):796-806. doi: 10.1016/S0140-6736(09)60918-1. Epub 2009 Aug 3. PMID 19647866
- [Result] DeJesus E, Rockstroh JK, Lennox JL, Saag MS, Lazzarin A, Zhao J, Wan H, Rodgers AJ, Walker ML, Miller M, DiNubile MJ, Nguyen BY, Teppler H, Leavitt R, Sklar P; STARTMRK Investigators. Efficacy of raltegravir versus efavirenz when combined with tenofovir/emtricitabine in treatment-naive HIV-1-infected patients: week-192 overall and subgroup analyses from STARTMRK. HIV Clin Trials. 2012 Jul-Aug;13(4):228-32. doi: 10.1310/hct1304-228. PMID 22849964
- [Result] Rockstroh JK, Lennox JL, Dejesus E, Saag MS, Lazzarin A, Wan H, Walker ML, Xu X, Zhao J, Teppler H, Dinubile MJ, Rodgers AJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK Investigators. Long-term treatment with raltegravir or efavirenz combined with tenofovir/emtricitabine for treatment-naive human immunodeficiency virus-1-infected patients: 156-week results from STARTMRK. Clin Infect Dis. 2011 Oct;53(8):807-16. doi: 10.1093/cid/cir510. PMID 21921224
- [Result] Rockstroh J, Teppler H, Zhao J, Sklar P, Harvey C, Strohmaier K, Leavitt R, Nguyen BY. Safety and efficacy of raltegravir in patients with HIV-1 and hepatitis B and/or C virus coinfection. HIV Med. 2012 Feb;13(2):127-31. doi: 10.1111/j.1468-1293.2011.00933.x. Epub 2011 May 22. PMID 21599819
- [Result] Rockstroh JK, Teppler H, Zhao J, Sklar P, Miller MD, Harvey CM, Strohmaier KM, Leavitt RY, Nguyen BY. Clinical efficacy of raltegravir against B and non-B subtype HIV-1 in phase III clinical studies. AIDS. 2011 Jul 17;25(11):1365-9. doi: 10.1097/QAD.0b013e328348065a. PMID 21522004
- [Result] Nguyen BY, Isaacs RD, Teppler H, Leavitt RY, Sklar P, Iwamoto M, Wenning LA, Miller MD, Chen J, Kemp R, Xu W, Fromtling RA, Vacca JP, Young SD, Rowley M, Lower MW, Gottesdiener KM, Hazuda DJ. Raltegravir: the first HIV-1 integrase strand transfer inhibitor in the HIV armamentarium. Ann N Y Acad Sci. 2011 Mar;1222:83-9. doi: 10.1111/j.1749-6632.2011.05972.x. PMID 21434946
- [Result] Teppler H, Brown DD, Leavitt RY, Sklar P, Wan H, Xu X, Lievano F, Lehman HP, Mast TC, Nguyen BY. Long-term safety from the raltegravir clinical development program. Curr HIV Res. 2011 Jan;9(1):40-53. doi: 10.2174/157016211794582650. PMID 21198432
- [Result] Lennox JL, Dejesus E, Berger DS, Lazzarin A, Pollard RB, Ramalho Madruga JV, Zhao J, Wan H, Gilbert CL, Teppler H, Rodgers AJ, Barnard RJ, Miller MD, Dinubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK Investigators. Raltegravir versus Efavirenz regimens in treatment-naive HIV-1-infected patients: 96-week efficacy, durability, subgroup, safety, and metabolic analyses. J Acquir Immune Defic Syndr. 2010 Sep;55(1):39-48. doi: 10.1097/QAI.0b013e3181da1287. PMID 20404738

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary therapy period: 14-Sep-2006 to 06-May-2009
  Multicenter (67) in the United States (18) and Ex-US (49)
Period: Overall Study
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Started | 282 | 284
Treated | 281 | 282
Completed | 210 | 184
Not Completed | 72 | 100
Not completed — Never Treated | 1 | 2
Not completed — Adverse Event | 14 | 28
Not completed — Lack of Efficacy | 6 | 10
Not completed — Lost to Follow-up | 12 | 22
Not completed — Protocol Violation | 5 | 3
Not completed — Withdrawal by Subject | 5 | 18
Not completed — Pregnancy | 4 | 2
Not completed — Completed, Did Not Enter Extension | 5 | 6
Not completed — Moved | 11 | 5
Not completed — Treatment with Prohibited Medication | 3 | 1
Not completed — Employment Interfered with Study Visits | 1 | 0
Not completed — Study Site Terminated | 2 | 0
Not completed — Miscellaneous | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s. | Total
Number analyzed (Participants) | 281 | 282 | 563
Age, Continuous [Mean (Full Range); unit: years] | 38 [19 to 67] | 37 [19 to 71] | 37 [19 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 51 | 105
  Male | 227 | 231 | 458
Race/Ethnicity, Customized [Number; unit: participants]
  White | 116 | 123 | 239
  Black | 33 | 23 | 56
  Asian | 36 | 32 | 68
  Hispanic | 60 | 67 | 127
  Others | 36 | 37 | 73
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Full Range); unit: Cells/mm^3] | 219 [1 to 620] | 217 [4 to 807] | 218 [1 to 807]
Plasma Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) [Geometric Mean (Full Range); unit: Copies/mL] | 103205 [400 to 750000] | 106215 [4410 to 750000] | 104702 [400 to 750000]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) <50 Copies/mL at Week 48
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <50 copies/mL at Week 48.
Time Frame: 48 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 280 | 281
Participants | 241 | 230

2. Secondary Outcome: Number of Participants Who Achieved HIV RNA <400 Copies/mL at Week 48
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <400 copies/mL at Week 48.
Time Frame: 48 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 280 | 281
Participants | 252 | 241

3. Secondary Outcome: Change From Baseline in Cluster of Differentiation Antigen 4 (CD4) Cell Count at Week 48
Description: Mean change from baseline at Week 48 in CD4 cell count (cells/mm3)
Time Frame: Baseline and Week 48
Population: Observed failure approach assuming baseline-carry-forward for all failures, exclude other missing values. Baseline CD4 cell count (cells/mm3) was carried forward for participants who discontinued assigned therapy due to lack of efficacy.
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm3)
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 258 | 251
CD4 Cell Count (cells/mm3) | 189.1 [173.9 to 204.3] | 163.3 [148.2 to 178.4]

4. Secondary Outcome: Number of Participants Who Achieved HIV RNA <50 Copies/mL at Week 96
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <50 copies/mL at Week 96.
Time Frame: 96 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants | 228 | 222

5. Secondary Outcome: Number of Participants Who Achieved HIV RNA <400 Copies/mL at Week 96
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <400 copies/mL at Week 96.
Time Frame: 96 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants | 240 | 229

6. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Description: Mean change from baseline at Week 96 in CD4 cell count (cells/mm3)
Time Frame: Baseline and Week 96
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm3)
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 249 | 243
CD4 Cell Count (cells/mm3) | 239.6 [219.8 to 259.4] | 224.8 [205.8 to 243.9]

7. Secondary Outcome: Number of Participants Who Achieved HIV RNA <50 Copies/mL at Week 156
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <50 copies/mL at Week 156.
Time Frame: 156 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants | 212 | 192

8. Secondary Outcome: Number of Participants Who Achieved HIV RNA <400 Copies/mL at Week 156
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <400 copies/mL at Week 156.
Time Frame: 156 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants | 224 | 203

9. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 156
Description: Mean change from baseline at Week 156 in CD4 cell count (cells/mm3)
Time Frame: Baseline and Week 156
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm3)
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 236 | 226
CD4 Cell Count (cells/mm3) | 331.7 [309.3 to 354.2] | 295.2 [271.3 to 319.0]

10. Secondary Outcome: Number of Participants Who Achieved HIV RNA <50 Copies/mL at Week 240
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <50 copies/mL at Week 240.
Time Frame: 240 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 279 | 279
Participants | 198 | 171

11. Secondary Outcome: Number of Participants Who Achieved HIV RNA <400 Copies/mL at Week 240
Description: Antiretroviral activity was evaluated for participants who achieved HIV RNA level <400 copies/mL at Week 240.
Time Frame: 240 Weeks
Population: All participants who took study medication and had HIV RNA tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 279 | 279
Participants | 206 | 181

12. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 240
Description: Mean change from baseline at Week 240 in CD4 cell count (cells/mm3)
Time Frame: Baseline and Week 240
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: CD4 Cell Count (cells/mm3)
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 222 | 212
CD4 Cell Count (cells/mm3) | 373.7 [344.6 to 402.8] | 311.6 [283.9 to 339.4]

13. Secondary Outcome: Number of Participants With Nervous System Symptoms Assessed by Review of Accumulated Safety Data up to Week 8
Description: Participants with dizziness, insomnia, somnolence, concentration impaired, depression, nightmare, confusional state, suicidal ideation, nervous system disorder, psychotic disorder, abnormal dreams, suicide attempt, acute psychosis, delirium, depressed level of consciousness, hallucination, auditory hallucination, completed suicide, and major depression
Time Frame: 8 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Nervous System Symptoms | 57 | 147
  Without Nervous System Symptoms | 224 | 135

14. Secondary Outcome: Number of Participants With CAEs at Week 96
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With CAEs | 265 | 274
  Without CAEs | 16 | 8

15. Secondary Outcome: Number of Participants With CAEs at Week 156
Description: as for outcome 14
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With CAEs | 267 | 276
  Without CAEs | 14 | 6

16. Secondary Outcome: Number of Participants With CAEs at Week 240
Description: as for outcome 14
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With CAEs | 271 | 276
  Without CAEs | 10 | 6

17. Secondary Outcome: Number of Participants With Serious CAEs at Week 96
Description: Serious CAEs are any AEs occurring at any dose that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose.
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious CAEs | 37 | 33
  Without Serious CAEs | 244 | 249

18. Secondary Outcome: Number of Participants With Serious CAEs at Week 156
Description: as for outcome 17
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious CAEs | 46 | 46
  Without Serious CAEs | 235 | 236

19. Secondary Outcome: Number of Participants With Serious CAEs at Week 240
Description: as for outcome 17
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious CAEs | 57 | 57
  Without Serious CAEs | 224 | 225

20. Secondary Outcome: Number of Participants With Drug-related CAEs at Week 96
Description: Adverse experiences (AEs) in this study were defined as "drug-related" if the investigator, who is a qualified physician, considered the AE as possibly, probably, or definitely related to MK-0518 or efavirenz alone or in combination with TRUVADA® or to TRUVADA® alone according to his/her best clinical judgment.
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With drug-related CAEs | 132 | 220
  Without drug-related CAEs | 149 | 62

21. Primary Outcome: Number of Participants With Clinical Adverse Experiences (CAEs) at Week 48
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study drug, whether or not considered related to the use of the product.
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Groups:
- MK-0518 400 mg b.i.d.: MK-0518 400 mg, which can be taken by mouth (PO) twice a day (b.i.d.) without regard to food, and placebo to efavirenz, which will be taken PO (q.h.s.) on an empty stomach preferably at bedtime. All participants will take one tablet of TRUVADA® (200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate) with food, daily with the morning dose of MK-0518. Dosing interval adjustment of TRUVADA® is recommended in all participants with creatinine clearance 30-49 mL/min.
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With CAEs | 253 | 272
  Without CAEs | 28 | 10

22. Primary Outcome: Number of Participants With Serious CAEs at Week 48
Description: as for outcome 17
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious CAEs | 28 | 27
  Without Serious CAEs | 253 | 255

23. Primary Outcome: Number of Participants With Drug-related CAEs at Week 48
Description: as for outcome 20
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Drug-related CAEs | 124 | 217
  Without Drug-related CAEs | 157 | 65

24. Primary Outcome: Number of Participants With Serious Drug-related CAEs at Week 48
Description: Serious CAEs are any AEs occurring at any dose that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose.
  Adverse experiences (AEs) in this study were defined as "drug-related" if the investigator, who is a qualified physician, considered the AE as possibly, probably, or definitely related to MK-0518 or efavirenz alone or in combination with TRUVADA® or to TRUVADA® alone according to his/her best clinical judgment.
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related CAEs | 4 | 5
  Without Serious Drug-related CAEs | 277 | 277

25. Primary Outcome: Number of Participants That Died by Week 48
Description: All participant deaths in the span of 48 weeks on study were recorded.
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Died | 2 | 0
  Did Not Die | 279 | 282

26. Primary Outcome: Number of Participants That Discontinued With CAEs at Week 48
Description: as for outcome 21
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued with CAEs | 9 | 17
  Did Not Discontinue with CAEs | 272 | 265

27. Primary Outcome: Number of Participants That Discontinued With Serious CAEs at Week 48
Description: as for outcome 17
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued with Serious CAEs | 7 | 4
  Did Not Discontinue with Serious CAEs | 274 | 278

28. Primary Outcome: Number of Participants That Discontinued With Drug-related CAEs at Week 48
Description: as for outcome 20
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued with Drug-related CAEs | 3 | 11
  Did not Discontinue with Drug-related CAEs | 278 | 271

29. Primary Outcome: Number of Participants That Discontinued With Serious Drug-related CAEs at Week 48
Description: as for outcome 24
Time Frame: 48 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontiued with Serious Drug-related CAEs | 1 | 2
  Did Not Discontinue with Serious Drug-related CAEs | 280 | 280

30. Primary Outcome: Number of Participants With Laboratory Adverse Experiences (LAEs) at Week 48
Description: A laboratory AE is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product.
Time Frame: 48 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With LAEs | 27 | 41
  Without LAEs | 254 | 241

31. Primary Outcome: Number of Participants With Serious LAEs at Week 48
Description: A laboratory AE is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product.
  Serious AEs are any AEs occurring at any dose that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose.
Time Frame: 48 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious LAEs | 0 | 1
  Without Serious LAEs | 281 | 281

32. Primary Outcome: Number of Participants With Drug-related LAEs at Week 48
Description: A laboratory AE is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product.
  Adverse experiences (AEs) in this study were defined as "drug-related" if the investigator, who is a qualified physician, considered the AE as possibly, probably, or definitely related to MK-0518 or efavirenz alone or in combination with TRUVADA® or to TRUVADA® alone according to his/her best clinical judgment.
Time Frame: 48 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Drug-related LAEs | 14 | 24
  Without Drug-related LAEs | 267 | 258

33. Primary Outcome: Number of Participants With Serious Drug-related LAEs at Week 48
Description: A laboratory AE is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product.
  Serious AEs are any AEs occurring at any dose that: results in death; or is life threatening; or results in a persistent or significant disability/incapacity; or results in or prolongs an existing inpatient hospitalization; or is a congenital anomaly/birth defect; or is a cancer; or is an overdose.
  Adverse experiences (AEs) in this study were defined as "drug-related" if the investigator, who is a qualified physician, considered the AE as possibly, probably, or definitely related to MK-0518 or efavirenz alone or in combination with TRUVADA® or to TRUVADA® alone according to his/her best clinical judgment.
Time Frame: 48 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related LAEs | 0 | 0
  Without Serious Drug-related LAEs | 281 | 282

34. Primary Outcome: Number of Participants Discontinued With LAEs at Week 48
Description: as for outcome 30
Time Frame: 48 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued with LAEs | 0 | 1
  Did Not Discontinue with LAEs | 281 | 281

35. Primary Outcome: Number of Participants Discontinued With Drug-related LAEs at Week 48
Description: A laboratory AE is defined as any unfavorable and unintended change in the chemistry of the body temporally associated with the use of the study product, whether or not considered related to the use of the product.
  Adverse events (AEs) in this study were defined as "drug-related" if the investigator considered the AE as possibly, probably, or definitely related to MK-0518 or efavirenz alone or in combination with TRUVADA® or to TRUVADA® alone.
Time Frame: 48 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued with Drug-related LAEs | 0 | 1
  Did Not Discontinue with Drug-related LAEs | 281 | 281

36. Secondary Outcome: Number of Participants With Drug-related CAEs at Week 156
Description: as for outcome 20
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With drug-related CAEs | 139 | 225
  Without drug-related CAEs | 142 | 57

37. Secondary Outcome: Number of Participants With Drug-related CAEs at Week 240
Description: as for outcome 20
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With drug-related CAEs | 146 | 226
  Without drug-related CAEs | 135 | 56

38. Secondary Outcome: Number of Participants With Serious Drug-related CAEs at Week 96
Description: as for outcome 24
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related CAEs | 6 | 5
  Without Serious Drug-related CAEs | 275 | 277

39. Secondary Outcome: Number of Participants With Serious Drug-related CAEs at Week 156
Description: as for outcome 24
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related CAEs | 6 | 6
  Without Serious Drug-related CAEs | 275 | 276

40. Secondary Outcome: Number of Participants With Serious Drug-related CAEs at Week 240
Description: as for outcome 24
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related CAEs | 8 | 7
  Without Serious Drug-related CAEs | 273 | 275

41. Secondary Outcome: Number of Participants That Died by Week 96
Description: All participant deaths in the span of 96 weeks on study were recorded.
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Died | 3 | 0
  Did Not Die | 278 | 282

42. Secondary Outcome: Number of Participants That Died by Week 156
Description: All participant deaths in the span of 156 weeks on study were recorded.
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Died | 4 | 1
  Did Not Die | 277 | 281

43. Secondary Outcome: Number of Participants That Died by Week 240
Description: All participant deaths in the span of 240 weeks on study were recorded.
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Died | 5 | 5
  Did Not Die | 276 | 277

44. Secondary Outcome: Number of Participants That Discontinued With CAEs at Week 96
Description: as for outcome 14
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With CAEs | 10 | 17
  Did Not Discontinue With CAEs | 271 | 265

45. Secondary Outcome: Number of Participants That Discontinued With CAEs at Week 156
Description: as for outcome 14
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With CAEs | 13 | 21
  Did Not Discontinue With CAEs | 268 | 261

46. Secondary Outcome: Number of Participants That Discontinued With CAEs at Week 240
Description: as for outcome 14
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With CAEs | 14 | 25
  Did Not Discontinue With CAEs | 267 | 257

47. Secondary Outcome: Number of Participants That Discontinued With Drug-related CAEs at Week 96
Description: as for outcome 20
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Drug-Related CAEs | 3 | 12
  Did Not Discontinue With Drug-Related CAEs | 278 | 270

48. Secondary Outcome: Number of Participants That Discontinued With Drug-related CAEs at Week 156
Description: as for outcome 20
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Drug-related CAEs | 3 | 14
  Did Not Discontinue With Drug-related CAEs | 278 | 268

49. Secondary Outcome: Number of Participants That Discontinued With Drug-related CAEs at Week 240
Description: as for outcome 20
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Drug-related CAEs | 3 | 14
  Did Not Discontinue With Drug-related CAEs | 278 | 268

50. Secondary Outcome: Number of Participants That Discontinued With Serious CAEs at Week 96
Description: as for outcome 17
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Serious CAEs | 8 | 5
  Did Not Discontinue With Serious CAEs | 273 | 277

51. Secondary Outcome: Number of Participants That Discontinued With Serious CAEs at Week 156
Description: as for outcome 17
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Serious CAEs | 10 | 6
  Did Not Discontinue With Serious CAEs | 271 | 276

52. Secondary Outcome: Number of Participants That Discontinued With Serious CAEs at Week 240
Description: as for outcome 17
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Serious CAEs | 11 | 10
  Did Not Discontinue With Serious CAEs | 270 | 272

53. Secondary Outcome: Number of Participants That Discontinued With Serious Drug-related CAEs at Week 96
Description: as for outcome 24
Time Frame: 96 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Serious Drug-related CAEs | 1 | 2
  Did Not Discontinue With Serious Drug-related CAEs | 280 | 280

54. Secondary Outcome: Number of Participants That Discontinued With Serious Drug-related CAEs at Week 156
Description: as for outcome 24
Time Frame: 156 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Serious Drug-related CAEs | 1 | 2
  Did Not Discontinue With Serious Drug-related CAEs | 280 | 280

55. Secondary Outcome: Number of Participants That Discontinued With Serious Drug-related CAEs at Week 240
Description: as for outcome 24
Time Frame: 240 Weeks
Population: All participants who took study medication were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Serious Drug-related CAEs | 1 | 2
  Did Not Discontinue With Serious Drug-related CAEs | 280 | 280

56. Secondary Outcome: Number of Participants With LAEs at Week 96
Description: as for outcome 30
Time Frame: 96 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With LAEs | 33 | 53
  Without LAEs | 248 | 229

57. Secondary Outcome: Number of Participants With LAEs at Week 156
Description: as for outcome 30
Time Frame: 156 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With LAEs | 41 | 63
  Without LAEs | 240 | 219

58. Secondary Outcome: Number of Participants With LAEs at Week 240
Description: as for outcome 30
Time Frame: 240 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With LAEs | 56 | 77
  Without LAEs | 225 | 205

59. Secondary Outcome: Number of Participants With Drug-related LAEs at Week 96
Description: as for outcome 32
Time Frame: 96 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Drug-related LAEs | 18 | 29
  Without Drug-related LAEs | 263 | 253

60. Secondary Outcome: Number of Participants With Drug-related LAEs at Week 156
Description: as for outcome 32
Time Frame: 156 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Drug-related LAEs | 22 | 33
  Without Drug-related LAEs | 259 | 249

61. Secondary Outcome: Number of Participants With Drug-related LAEs at Week 240
Description: as for outcome 32
Time Frame: 240 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Drug-related LAEs | 26 | 43
  Without Drug-related LAEs | 255 | 239

62. Secondary Outcome: Number of Participants With Serious LAEs at Week 96
Description: as for outcome 31
Time Frame: 96 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious LAEs | 0 | 1
  Without Serious LAEs | 281 | 281

63. Secondary Outcome: Number of Participants With Serious LAEs at Week 156
Description: as for outcome 31
Time Frame: 156 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious LAEs | 0 | 2
  Without Serious LAEs | 281 | 280

64. Secondary Outcome: Number of Participants With Serious LAEs at Week 240
Description: as for outcome 31
Time Frame: 240 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious LAEs | 0 | 2
  Without Serious LAEs | 281 | 280

65. Secondary Outcome: Number of Participants With Serious Drug-related LAEs at Week 96
Description: as for outcome 33
Time Frame: 96 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related CAEs | 0 | 0
  Without Serious Drug-related CAEs | 281 | 282

66. Secondary Outcome: Number of Participants With Serious Drug-related LAEs at Week 156
Description: as for outcome 33
Time Frame: 156 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related CAEs | 0 | 1
  Without Serious Drug-related CAEs | 281 | 281

67. Secondary Outcome: Number of Participants With Serious Drug-related LAEs at Week 240
Description: as for outcome 33
Time Frame: 240 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  With Serious Drug-related LAEs | 0 | 1
  Without Serious Drug-related LAEs | 281 | 281

68. Secondary Outcome: Number of Participants Discontinued With LAEs at Week 96
Description: as for outcome 30
Time Frame: 96 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With LAEs | 0 | 2
  Did Not Discontinue With LAEs | 281 | 280

69. Secondary Outcome: Number of Participants Discontinued With LAEs at Week 156
Description: as for outcome 30
Time Frame: 156 Weeks
Population: All patients who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With LAEs | 0 | 3
  Did Not Discontinue With LAEs | 281 | 279

70. Secondary Outcome: Number of Participants Discontinued With LAEs at Week 240
Description: as for outcome 30
Time Frame: 240 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With LAEs | 0 | 3
  Did Not Discontinue With LAEs | 281 | 279

71. Secondary Outcome: Number of Participants Discontinued With Drug-related LAEs at Week 96
Description: as for outcome 32
Time Frame: 96 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Drug-related LAEs | 0 | 1
  Did Not Discontinue With Drug-related LAEs | 281 | 281

72. Secondary Outcome: Number of Participants Discontinued With Drug-related LAEs at Week 156
Description: as for outcome 32
Time Frame: 156 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Drug-related LAEs | 0 | 2
  Did Not Discontinue With Drug-related LAEs | 281 | 280

73. Secondary Outcome: Number of Participants Discontinued With Drug-related LAEs at Week 240
Description: as for outcome 32
Time Frame: 240 Weeks
Population: All participants who took study medication and had any laboratory tests performed were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Number analyzed (Participants) | 281 | 282
Participants
  Discontinued With Drug-related LAEs | 0 | 2
  Did Not Discontinue With Drug-related LAEs | 281 | 280

ADVERSE EVENTS:
Time Frame: 240 weeks
Description: Adverse events are reported for the entire 240-week study.
Groups:
- MK-0518 400 mg b.i.d.: MK-0518 400 mg taken by mouth (PO) twice a day (b.i.d.) without regard to food, and placebo to efavirenz, taken PO (q.h.s.) on an empty stomach preferably at bedtime (q.h.s.). All participants will take one tablet of TRUVADA® (200 mg of emtricitabine and 300 mg of tenofovir disoproxil fumarate) daily with food with the morning dose of MK-0518. Dosing interval adjustment of TRUVADA® is recommended in all participants with creatinine clearance 30-49 mL/min.
- Efavirenz 600 mg q.h.s.: Efavirenz 600 mg taken by mouth on an empty stomach preferably at bedtime (q.h.s.), and placebo to MK-0518 taken PO twice a day (b.i.d.) without regard to food. All participants will take one tablet of TRUVADA® with food, daily with the morning dose of placebo. Dosing interval adjustment of TRUVADA® is recommended in all participants with creatinine clearance 30-49 mL/min.
Arm/Group | MK-0518 400 mg b.i.d. | Efavirenz 600 mg q.h.s.
Serious Adverse Events (participants affected / at risk) | 57/281 | 59/282
Other Adverse Events (participants affected / at risk) | 257/281 | 263/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0518 400 mg b.i.d. (N=281) | Efavirenz 600 mg q.h.s. (N=282)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Branchial cleft cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Heart disease congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Immune reconstitution syndrome (Immune system disorders) | 5 (5) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 3 (3)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bone tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (2)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 2 (2) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 1 (1) | 0 (0)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Secondary syphilis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (2)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Accidental exposure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 3 (3)
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Kaposi's sarcoma AIDS related (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 6 (7)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (6) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 3 (6) | 3 (3)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Mental disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Psychosomatic disease (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 4 (4) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arteriosclerosis obliterans (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0518 400 mg b.i.d. (N=281) | Efavirenz 600 mg q.h.s. (N=282)
Abdominal pain (Gastrointestinal disorders) | 24 (30) | 19 (23)
Abdominal pain upper (Gastrointestinal disorders) | 8 (16) | 19 (20)
Diarrhoea (Gastrointestinal disorders) | 72 (104) | 76 (105)
Dyspepsia (Gastrointestinal disorders) | 25 (27) | 14 (18)
Flatulence (Gastrointestinal disorders) | 14 (17) | 19 (19)
Nausea (Gastrointestinal disorders) | 47 (68) | 41 (52)
Vomiting (Gastrointestinal disorders) | 23 (29) | 30 (38)
Asthenia (General disorders) | 17 (24) | 16 (16)
Fatigue (General disorders) | 26 (29) | 38 (46)
Pyrexia (General disorders) | 44 (62) | 39 (50)
Bronchitis (Infections and infestations) | 29 (48) | 30 (48)
Gastroenteritis (Infections and infestations) | 17 (19) | 19 (20)
Genital herpes (Infections and infestations) | 12 (17) | 15 (19)
Herpes zoster (Infections and infestations) | 14 (17) | 16 (19)
Influenza (Infections and infestations) | 33 (58) | 38 (68)
Nasopharyngitis (Infections and infestations) | 75 (121) | 63 (123)
Pharyngitis (Infections and infestations) | 27 (33) | 26 (33)
Sinusitis (Infections and infestations) | 23 (31) | 23 (31)
Upper respiratory tract infection (Infections and infestations) | 60 (95) | 57 (85)
Alanine aminotransferase increased (Investigations) | 19 (33) | 28 (49)
Aspartate aminotransferase increased (Investigations) | 21 (37) | 25 (44)
Decreased appetite (Metabolism and nutrition disorders) | 12 (18) | 19 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (29) | 33 (34)
Back pain (Musculoskeletal and connective tissue disorders) | 34 (43) | 28 (34)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12) | 15 (19)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (23) | 15 (17)
Dizziness (Nervous system disorders) | 46 (49) | 108 (140)
Headache (Nervous system disorders) | 73 (127) | 80 (109)
Somnolence (Nervous system disorders) | 3 (5) | 22 (27)
Abnormal dreams (Psychiatric disorders) | 23 (29) | 37 (43)
Anxiety (Psychiatric disorders) | 25 (25) | 31 (31)
Depression (Psychiatric disorders) | 27 (32) | 33 (38)
Insomnia (Psychiatric disorders) | 44 (56) | 42 (49)
Nightmare (Psychiatric disorders) | 10 (12) | 15 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (64) | 34 (47)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 22 (22) | 15 (15)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 6 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (12) | 15 (15)
Rash (Skin and subcutaneous tissue disorders) | 22 (26) | 39 (46)
Hypertension (Vascular disorders) | 18 (20) | 18 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.